CLINICAL TRIAL: NCT03941106
Title: A Pilot Study of Intermittent Accelerated Burst Transcranial Magnetic Stimulation (aTBS) to Treat Depression: a Randomized, Single-blind, Delayed-start Trial
Brief Title: Accelerated Transcranial Magnetic Stimulation (aTBS) to Treat Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CNIG18may-0001
Record Dates: First submitted 2019-04-07; First posted 2019-05-07 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2021-08

CONDITIONS: Depression
Keywords: rTMS, depression, accelerated
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left aTMS (Experimental)
  Interventions: Device: Accelerated repetitive transcranial magnetic stimulation
- Right aTMS (Experimental)
  Interventions: Device: Accelerated repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Accelerated repetitive transcranial magnetic stimulation — Subjects will be given accelerated left sided rTMS and randomized to more of the same accelerated rTMS if not meeting remission criteria for depression or a different type of rTMS on the right side

SUMMARY:
The primary aims of this study are to investigate the efficacy of L DLPFC accelerated TMS (aTMS) in patients with depression in Singapore and to assess the whether a 1-week course of treatment is as effective as a 4-week course of non-accelerated treatment and if additional aTMS or different aTMS treatments will be more efficacious in non-responders to initial aTMS treatment.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (TMS) is a technique for stimulating brain activity using transient magnetic field to induce an electrical current in the brain producing firing of focal groups of brain cells. TMS is beginning to emerge in routine clinical practice as a treatment for depression. The predominant hypothesis is that depressed patients benefit from left sided high-frequency TMS (LHF-TMS) over the left dorsolateral prefrontal cortex (DLPFC)(1). A major limitation of rTMS is the large amount of time taken for a standard protocol (38 minutes a day for 20-30 working days). The optimal type and duration of TMS is still uncertain , as is the optimal strategy for continuing or changing type of rTMS if there is poor initial response.(1) One potential strategy to improve the acceptability of rTMS is to compress or accelerate the administration of rTMS (aTMS) by administering multiple sessions of rTMS over a shorter period of time to have equivalent efficacy in shorter period of time. Various studies of aTMS (2-9) have been safely conducted with anywhere from 2 (3) to 10 (2) sessions of rTMS a day for a total of 9 (5) - 20 (4, 7) sessions of TMS over 2 (2) to 9 (8) days. These studies showed that aTMS was safe and efficacious, with no significant side effects reported and a high level of patient acceptability and significant improvements in subjects' depression after the aTMS. However, there is no data on whether subjects who do not response to aTMS will benefit from more of the same TMS or from changing the mode of rTMS. The only study investigating this issue investigated normal rTMS, not aTMS, and did not find a significant difference in response to different forms of rTMS in initial non-responders (10). Our own observations and some preliminary evidence suggest that there may be a delayed response to TMS in some patients (11, 12). Thus, instead of the usual practice of giving 4-6 weeks stimulation (every weekday) and assessing for response at the end of the stimulation period, the same outcome may be achieved by giving a shorter period of stimulation (eg 1 weeks), waiting 2-4 weeks, then assessing response and the need for further TMS treatment. Further, giving more than 1 treatment per day has been shown to be effective (13) and may lead to more efficient treatment, i.e. fewer days to response and less requirement for patient attendance at the treatment centre (2-9).

This pilot study will contribute to existing knowledge by being possibly the first group in South East Asia to investigate the immediate and delayed efficacy of aTMS in the local population (i.e. in an Asian setting) as well as whether continuing or changing the type of rTMS is more efficacious in subjects who do not respond to initial aTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years.
2. DSM-V diagnosis of current Major Depressive Episode.
3. Montgomery-Asberg Depression Rating Scale score of 20 or more.
4. Able to give informed consent.

Exclusion Criteria:

1. DSM-V psychotic disorder.
2. Drug or alcohol abuse or dependence (preceding 3 months).
3. Inadequate response to ECT (current episode of depression).
4. Rapid clinical response required, e.g. high suicide risk.
5. Significant neurological disorder, which may pose increased risks with TMS, e.g., epilepsy.
6. Metal in the cranium, skull defects, pacemaker, cochlear implant, medication pump or other electronic device.
7. Pregnancy.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Remission as assessed by The Montgomery-Åsberg Depression Rating Scale (MADRS) | 3 weeks
  The MADRS is a 0-60 point scale to measure depression severity with a higher number indicating more severe depression. Remission from depression is defined as 10 or less. Moderate to severe depression is defined as 20 or more.

SECONDARY OUTCOMES:
Remission as assessed by The Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 weeks
  A MADRS score of 10 or less.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tor PC, Galvez V, Goldstein J, George D, Loo CK. Pilot Study of Accelerated Low-Frequency Right-Sided Transcranial Magnetic Stimulation for Treatment-Resistant Depression. J ECT. 2016 Sep;32(3):180-2. doi: 10.1097/YCT.0000000000000306. PMID 26909825
- [Derived] Tan XW, Abdin E, Tor PC. Accelerated transcranial magnetic stimulation (aTMS) to treat depression with treatment switching: study protocol of a pilot, randomized, delayed-start trial. Pilot Feasibility Stud. 2021 May 5;7(1):104. doi: 10.1186/s40814-021-00845-9. PMID 33952345